CLINICAL TRIAL: NCT01515189
Title: A Randomized Double-Blind Phase III Study of Ipilimumab Administered at 3 mg/kg Versus at 10 mg /kg in Subjects With Previously Treated or Untreated Unresectable or Metastatic Melanoma
Brief Title: Phase 3 Trial in Subjects With Metastatic Melanoma Comparing 3 mg/kg Ipilimumab Versus 10 mg/kg Ipilimumab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA184-169; 2011-004029-28 (EudraCT Number)
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Results first posted 2017-03-24 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Ipilimumab (3 mg/kg) (Experimental): Ipilimumab 3 mg/kg solution intravenously once every 3 weeks for 4 doses; option for Re-induction, until disease progression or unacceptable toxicity
  Interventions: Biological: Ipilimumab
- Arm 2: Ipilimumab (10 mg/kg) (Experimental): Ipilimumab 10 mg/kg solution intravenously once every 3 weeks for 4 doses; option for Re-induction, until disease progression or unacceptable toxicity
  Interventions: Biological: Ipilimumab

INTERVENTIONS:
Biological: Ipilimumab
  Other Names: Yervoy; BMS-734016

SUMMARY:
The purpose of this study is to determine whether giving Ipilimumab at a dose of 10mg/kg will extend the lives of subjects with unresectable or metastatic melanoma more than giving Ipilimumab at a dose of 3 mg/kg

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Unresectable Stage III or Stage IV melanoma
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Brain metastases with symptoms or requiring treatment
* History of autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 831 (Actual)
Dates: Start 2012-02-17 (Actual); Primary Completion 2016-02-06 (Actual); Study Completion 2017-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (87):
- United States (11):
  - The Angeles Clinic And Research Institute, Los Angeles, California
  - University Of California Los Angeles, Los Angeles, California
  - Baptist Cancer Institute, Jacksonville, Florida
  - Orlando Health, Inc, Orlando, Florida
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Providence Portland Medical Center, Portland, Oregon
  - St. Luke's Cancer Center - Anderson Campus, Easton, Pennsylvania
  - Seattle Cancer Care Alliance, Seattle, Washington
- Argentina (2):
  - Local Institution, San Miguel de Tucumán, Tucumán Province
  - Fundacion Cidea, Buenos Aires
- Australia (6):
  - Local Institution, Camperdown, New South Wales
  - Local Institution, Coffs Harbour, New South Wales
  - Local Institution, Brisbane, Queensland
  - Local Institution, Southport, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Heidelberg, Victoria
- Austria (2):
  - Local Institution, Linz
  - Local Institution, Vienna
- Belgium (2):
  - Local Institution, Brussels
  - Local Institution, Leuven
- Canada (3):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Halfax, Nova Scotia
  - Local Institution, Montreal, Quebec
- Czechia (3):
  - Local Institution, Brno
  - Local Institution, Olomouc
  - Local Institution, Prague
- Denmark (3):
  - Local Institution, Aarhus
  - Local Institution, Herlev
  - Local Institution, Odense
- France (11):
  - Local Institution, Bordeaux
  - Local Institution, Dijon
  - Local Institution, Grenoble
  - Local Institution, Lille
  - Local Institution, Marseille
  - Local Institution, Nantes
  - Local Institution, Paris
  - Local Institution, Pierre-Bénite
  - Local Institution, Reims
  - Local Institution, Toulouse
  - Local Institution, Villejuif
- Germany (8):
  - Local Institution, Buxtehude
  - Local Institution, Essen
  - Local Institution, Hanover
  - Local Institution, Heidelberg
  - Local Institution, Kiel
  - Local Institution, Mainz
  - Local Institution, Munich
  - Local Institution, Tübingen
- Hungary (3):
  - Local Institution, Budapest
  - Local Institution, Kaposvár
  - Local Institution, Szeged
- Local Institution, Jerusalem, Israel
- Italy (6):
  - Local Institution, Meldola (fc)
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Padua
  - Local Institution, Roma
  - Local Institution, Siena
- Local Institution, Leon, Guanajato, Guanajuato, Mexico
- Netherlands (3):
  - Local Institution, Amsterdam
  - Local Institution, Groningen
  - Local Institution, Leiden
- Norway (2):
  - Local Institution, Bergen
  - Local Institution, Oslo
- Poland (3):
  - Local Institution, Gdansk
  - Local Institution, Poznan
  - Local Institution, Warsaw
- South Africa (3):
  - Local Institution, Cape Town, Western Cape
  - Local Institution, George, Western Cape
  - Local Institution, Rondebosch, Western Cape
- Spain (5):
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Navarra
  - Instituto Valenciano De Oncologia, Valencia
  - Local Institution, Valencia
- Sweden (4):
  - Local Institution, Gothenberg
  - Local Institution, Lund
  - Local Institution, Stockholm
  - Local Institution, Umeå
- Local Institution, Lausanne, Switzerland
- United Kingdom (4):
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Glasgow, Scotland, Strathclyde
  - Local Institution, London
  - Local Institution, Swansea

REFERENCES:
- [Derived] Ascierto PA, Del Vecchio M, Mackiewicz A, Robert C, Chiarion-Sileni V, Arance A, Lebbe C, Svane IM, McNeil C, Rutkowski P, Loquai C, Mortier L, Hamid O, Bastholt L, Dreno B, Schadendorf D, Garbe C, Nyakas M, Grob JJ, Thomas L, Liszkay G, Smylie M, Hoeller C, Ferraresi V, Grange F, Gutzmer R, Pikiel J, Hosein F, Simsek B, Maio M. Overall survival at 5 years of follow-up in a phase III trial comparing ipilimumab 10 mg/kg with 3 mg/kg in patients with advanced melanoma. J Immunother Cancer. 2020 Jun;8(1):e000391. doi: 10.1136/jitc-2019-000391. PMID 32503946
- [Derived] Feng Y, Wang X, Suryawanshi S, Bello A, Roy A. Linking Tumor Growth Dynamics to Survival in Ipilimumab-Treated Patients With Advanced Melanoma Using Mixture Tumor Growth Dynamic Modeling. CPT Pharmacometrics Syst Pharmacol. 2019 Nov;8(11):825-834. doi: 10.1002/psp4.12454. Epub 2019 Aug 13. PMID 31334596
- [Derived] Ascierto PA, Del Vecchio M, Robert C, Mackiewicz A, Chiarion-Sileni V, Arance A, Lebbe C, Bastholt L, Hamid O, Rutkowski P, McNeil C, Garbe C, Loquai C, Dreno B, Thomas L, Grob JJ, Liszkay G, Nyakas M, Gutzmer R, Pikiel J, Grange F, Hoeller C, Ferraresi V, Smylie M, Schadendorf D, Mortier L, Svane IM, Hennicken D, Qureshi A, Maio M. Ipilimumab 10 mg/kg versus ipilimumab 3 mg/kg in patients with unresectable or metastatic melanoma: a randomised, double-blind, multicentre, phase 3 trial. Lancet Oncol. 2017 May;18(5):611-622. doi: 10.1016/S1470-2045(17)30231-0. Epub 2017 Mar 27. PMID 28359784
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 831 participants were enrolled; 727 were randomized to a treatment group; 726 received at least one dose of study treatment. Of the 105 participants not treated, 81 no longer met study criteria, 11 withdrew consent, 4 suffered an Adverse Event, 4 died, and 5 were not treated due to investigator decision or other reasons.
Groups:
- Ipilimumab (10 mg/kg): Ipilimumab 10 mg/kg solution intravenously once every 3 weeks for 4 doses or until disease progression or unacceptable toxicity
- Ipilimumab (3 mg/kg): Ipilimumab 3 mg/kg solution intravenously once every 3 weeks for 4 doses or until disease progression or unacceptable toxicity
Period: Induction
Arm/Group | Ipilimumab (10 mg/kg) | Ipilimumab (3 mg/kg)
Started | 365 (Includes 1 subject who was randomized but not treated due to an Adverse Event before treatment) | 362
Completed | 128 | 130
Not Completed | 237 | 232
Not completed — Disease Progression | 109 | 155
Not completed — Study drug toxicity | 86 | 36
Not completed — Death | 24 | 17
Not completed — Adverse Event | 14 | 9
Not completed — Withdrawal by Subject | 3 | 9
Not completed — No longer meets study criteria | 0 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 0 | 4
Period: First Re-Induction Phase
Arm/Group | Ipilimumab (10 mg/kg) | Ipilimumab (3 mg/kg)
Started | 23 | 32
Completed | 9 | 17
Not Completed | 14 | 15
Not completed — Disease progression | 6 | 14
Not completed — Study drug toxicity | 5 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — No longer meets study criteria | 1 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipilimumab (10 mg/kg) | Ipilimumab (3 mg/kg) | Total
Number analyzed (Participants) | 365 | 362 | 727
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 224 | 208 | 432
  >=65 years | 141 | 154 | 295
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (14.52) | 60.7 (13.22) | 59.7 (13.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 131 | 277
  Male | 219 | 231 | 450

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is defined for each participant as the time between randomization date and death due to any cause. The survival time for participants who had not died was censored at the last known alive date. Median and associated 2-sided 95% confidence intervals were calculated using the method of Brookmeyer and Crowley.
Time Frame: Approximately 48 months (assessed up to February 2016)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab (10 mg/kg) | Ipilimumab (3 mg/kg)
Number analyzed (Participants) | 365 | 362
months | 15.70 [11.63 to 17.84] | 11.53 [9.86 to 13.27]
Statistical Analysis 1: Comparison: Ipilimumab (10 mg/kg) vs Ipilimumab (3 mg/kg); Test type: Superiority; p = 0.0400, Log Rank — Analysis stratified by ECOG performance status (0 vs. 1), prior treatment for metastatic melanoma (yes vs. no) and M-stage (M0/M1a/M1b vs. M1c without brain metastases vs. M1c with brain metastases); Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.70 to 0.99] — Hazard of 10 mg/kg ipilimumab over hazard of 3 mg/kg, with 2-sided 95% confidence intervals are based on a Cox proportional hazards model

2. Secondary Outcome: Progression Free Survival (PFS) by mWHO Criteria
Description: PFS was defined as the time between randomization date and the date of progression or death, whichever occurred first. A participant who died without reported prior progression was considered to have progressed on the date of death. For a participant who underwent resection post randomization, PFS was censored on last tumor assessment date prior to resection. For those who remained alive and had not progressed, PFS was censored on last evaluable tumor assessment date. Participants who had not died and had no recorded post-baseline tumor assessment were censored at the day of randomization. For participants who had Progressive Disease (PD) prior to Week 12 and a subsequent assessment of Stable Disease (SD), Partial Response (PR), or Complete Response (CR), the date of PD following response was used in the analysis of PFS; otherwise these participants were censored on the date of their last tumor assessment. Median and 2-sided 95% CIs were calculated with Brookmeyer Crowley method.
Time Frame: From date of randomization until 540 death events occurred (approximately 48 months)
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab (10 mg/kg) | Ipilimumab (3 mg/kg)
Number analyzed (Participants) | 365 | 362
months | 2.83 [2.79 to 2.99] | 2.79 [2.76 to 2.83]
Statistical Analysis 1: Comparison: Ipilimumab (10 mg/kg) vs Ipilimumab (3 mg/kg); Test type: Superiority; p = 0.1548, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.76 to 1.04] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Best Overall Response Rate (BORR) by mWHO Criteria
Description: BORR by treatment arm was defined as the total number of randomized participants in the arm whose BOR is CR or PR, divided by the total number of randomized participants in the arm. Any participant who was unevaluable for BOR, e.g. on account of missing or "not evaluable" assessments, was included in the denominator of the calculation (i.e. was considered a non-responder with respect to the BORR endpoint). 95% 2-sided exact confidence intervals were computed using the method of Clopper and Pearson.
Time Frame: From date of randomization until 540 death events occurred (approximately 48 months)
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants with BORR
Arm/Group | Ipilimumab (10 mg/kg) | Ipilimumab (3 mg/kg)
Number analyzed (Participants) | 365 | 362
percentage of participants with BORR | 15.3 [11.8 to 19.5] | 12.2 [9.0 to 16.0]

4. Secondary Outcome: Disease Control Rate (DCR) by mWHO Criteria
Description: DCR by treatment arm was defined as the total number of randomized participants in the arm whose BOR is CR, PR or SD, divided by the total number of randomized participants in the arm. Any participant who was unevaluable for Disease Control (DC), (e.g. on account of missing or "not evaluable" assessments), was included in the denominator of the calculation (i.e. was considered a non-responder with respect to the DCR endpoint). 95% 2-sided exact confidence intervals were computed using the Clopper and Pearson method.
Time Frame: From date of randomization until 540 death events occurred (approximately 48 months)
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants with DC
Arm/Group | Ipilimumab (10 mg/kg) | Ipilimumab (3 mg/kg)
Number analyzed (Participants) | 365 | 362
percentage of participants with DC | 31.5 [26.8 to 36.5] | 27.9 [23.3 to 32.8]

5. Secondary Outcome: Duration of Response (DOR) by mWHO Criteria
Description: Duration of response for participants whose BOR was CR or PR was defined as the time between the date measurement criteria were first met for overall response of PR or CR (whichever status was recorded first) and the date of disease progression or death (whichever occurred first). For participants who underwent tumor resection following response but prior to disease progression, duration of response was censored on the date of last evaluable tumor assessment prior to resection. For participants who had BOR of SD, PR or CR at Week 12, or a confirmed response of PR or CR before Week 12, the date of PD following thereafter (where available) was used in the analysis of duration of response. For those participants who remained alive and had not progressed following response, duration of response was censored on the date of last evaluable tumor assessment. Median and associated 2-sided 95% confidence intervals were calculated using the Brookmeyer Crowley method.
Time Frame: From date of randomization until 540 death events occurred (approximately 48 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab (10 mg/kg) | Ipilimumab (3 mg/kg)
Number analyzed (Participants) | 365 | 362
months | 16.33 [5.98 to 23.98] | 15.90 [10.35 to NA] — The upper 95% CI for DOR was not reached.

6. Secondary Outcome: Duration of Stable Disease by mWHO Criteria
Description: Duration of stable disease was defined for participants whose BOR was SD as the time between when SD was first documented and the date of PD or death (whichever occurred first). For a participant who underwent tumor resection following Week 12 but prior to disease progression, duration of stable disease was censored on the date of the last evaluable tumor assessment prior to resection. For participants who had BOR of SD at Week 12, the date of PD following thereafter (where available) was used in the analysis of duration of stable disease. For participants with BOR of SD who had not subsequently progressed and who remained alive, duration of stable disease was censored on the date of last evaluable tumor assessment. Median and associated 2-sided 95% confidence intervals were calculated using the Brookmeyer and Crowley method.
Time Frame: From date of randomization until 540 death events occurred (approximately 48 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab (10 mg/kg) | Ipilimumab (3 mg/kg)
Number analyzed (Participants) | 365 | 362
months | 5.55 [3.02 to 8.02] | 3.19 [2.73 to 5.55]

7. Secondary Outcome: Rate of Overall Survival
Description: OS is defined for each participant as the time between randomization date and death due to any cause. The survival time for participants who had not died was censored at the last known alive date. Survival rates were calculated based on Kaplan-Meier estimation with log-log transformed confidence intervals. The survival rate at x year(s) is defined as the probability that a subject is alive at x year(s) following randomization.
Time Frame: Approximately 66 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ipilimumab (10 mg/kg) | Ipilimumab (3 mg/kg)
Number analyzed (Participants) | 365 | 362
percentage of participants
  Survival rate at 1 year | 54.28 [49.01 to 59.25] | 47.62 [42.35 to 52.70]
  Survival rate at 2 years | 38.46 [33.44 to 43.45] | 30.97 [26.21 to 35.84]
  Survival rate at 3 years | 31.16 [26.44 to 35.98] | 23.15 [18.88 to 27.69]
  Survival rate at 4 years | 26.63 [22.17 to 31.28] | 20.25 [16.21 to 24.62]
  Survival rate at 5 years | 24.90 [20.54 to 29.48] | 18.78 [14.87 to 23.05]

8. Secondary Outcome: Overall Survival of Participants With Brain Metastases at Baseline
Description: OS for each participant with brain metastases at baseline was measured as the time between randomization date and death due to any cause. The survival time for participants who had not died was censored at the last known alive date. Median OS, and associated 2-sided 95% confidence intervals were calculated using the Brookmeyer and Crowley method.
Time Frame: From date of randomization until 540 death events occurred (approximately 48 months)
Population: All randomized participants with brain metastases at baseline
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab (10 mg/kg) | Ipilimumab (3 mg/kg)
Number analyzed (Participants) | 65 | 62
months | 7.00 [3.98 to 12.78] | 5.67 [4.21 to 6.97]
Statistical Analysis 1: Comparison: Ipilimumab (10 mg/kg) vs Ipilimumab (3 mg/kg); Test type: Superiority; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.49 to 1.04] — Hazard of 10 mg/kg ipilimumab over hazard of 3 mg/kg. Based on an unstratified Cox proportional hazards model for subset of participants with brain metastases

ADVERSE EVENTS:
Time Frame: From Day 1 of study treatment until 90 days following last day of study treatment, up to study completion (August 2017)
Arm/Group | 10 MG/KG IPILIMUMAB | 3 MG/KG IPILIMUMAB
Serious Adverse Events (participants affected / at risk) | 245/364 | 194/362
Other Adverse Events (participants affected / at risk) | 319/364 | 302/362
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 MG/KG IPILIMUMAB (N=364) | 3 MG/KG IPILIMUMAB (N=362)
Anaemia (Blood and lymphatic system disorders) | 5 | 4
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2
Pericardial effusion (Cardiac disorders) | 1 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Carney complex (Congenital, familial and genetic disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 2 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 2 | 1
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 2 | 2
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Diabetes insipidus (Endocrine disorders) | 1 | 0
Endocrine disorder (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypophysitis (Endocrine disorders) | 16 | 9
Hypopituitarism (Endocrine disorders) | 5 | 3
Hypothalamo-pituitary disorder (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Lymphocytic hypophysitis (Endocrine disorders) | 1 | 2
Thyroiditis (Endocrine disorders) | 2 | 0
Thyrotoxic crisis (Endocrine disorders) | 0 | 1
Eye pain (Eye disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 2 | 3
Autoimmune colitis (Gastrointestinal disorders) | 4 | 4
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 33 | 13
Colitis ulcerative (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 42 | 22
Gastritis (Gastrointestinal disorders) | 3 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhagic ascites (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 2 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 3
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 3
Asthenia (General disorders) | 2 | 2
Chest pain (General disorders) | 1 | 2
Death (General disorders) | 1 | 0
Fatigue (General disorders) | 5 | 1
General physical health deterioration (General disorders) | 10 | 12
Generalised oedema (General disorders) | 0 | 1
Hyperthermia (General disorders) | 2 | 0
Influenza like illness (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Oedema (General disorders) | 1 | 0
Pain (General disorders) | 1 | 5
Performance status decreased (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 9 | 5
Ulcer haemorrhage (General disorders) | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 4 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 6 | 2
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 5 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 2 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Bartholinitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Cytomegalovirus colitis (Infections and infestations) | 1 | 1
Encephalitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 2 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Hepatitis viral (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 3 | 0
Liver abscess (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 2 | 0
Lymph node abscess (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pleural infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 4
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 2
Septic shock (Infections and infestations) | 2 | 2
Staphylococcal infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Viral infection (Infections and infestations) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Radiation dysphagia (Injury, poisoning and procedural complications) | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 6 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 1
Blood potassium increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Liver function test increased (Investigations) | 2 | 0
Transaminases increased (Investigations) | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 54 | 60
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Metastases to eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to muscle (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Neoplasm swelling (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Brain oedema (Nervous system disorders) | 1 | 0
Central nervous system haemorrhage (Nervous system disorders) | 2 | 0
Cerebellar haemorrhage (Nervous system disorders) | 1 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 1 | 0
Facial paresis (Nervous system disorders) | 1 | 0
Guillain-barre syndrome (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 5 | 2
Hemiparesis (Nervous system disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 0 | 1
Intensive care unit acquired weakness (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 3 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Neurological decompensation (Nervous system disorders) | 2 | 0
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 2
Sciatica (Nervous system disorders) | 1 | 1
Seizure (Nervous system disorders) | 1 | 2
Spinal cord compression (Nervous system disorders) | 2 | 2
Syncope (Nervous system disorders) | 3 | 1
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 2
Agitation (Psychiatric disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 3
Depressed mood (Psychiatric disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 3
Nephritis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 2
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Pulmonary microemboli (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2
Embolism (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 10 MG/KG IPILIMUMAB (N=364) | 3 MG/KG IPILIMUMAB (N=362)
Anaemia (Blood and lymphatic system disorders) | 24 | 17
Abdominal pain (Gastrointestinal disorders) | 33 | 34
Constipation (Gastrointestinal disorders) | 38 | 40
Diarrhoea (Gastrointestinal disorders) | 140 | 105
Nausea (Gastrointestinal disorders) | 59 | 74
Vomiting (Gastrointestinal disorders) | 43 | 34
Asthenia (General disorders) | 68 | 60
Fatigue (General disorders) | 86 | 95
Oedema peripheral (General disorders) | 25 | 22
Pyrexia (General disorders) | 59 | 43
Alanine aminotransferase increased (Investigations) | 27 | 12
Aspartate aminotransferase increased (Investigations) | 27 | 8
Weight decreased (Investigations) | 29 | 25
Decreased appetite (Metabolism and nutrition disorders) | 52 | 51
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 26
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 | 21
Dizziness (Nervous system disorders) | 16 | 22
Headache (Nervous system disorders) | 56 | 66
Insomnia (Psychiatric disorders) | 19 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 33 | 32
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 | 26
Pruritus (Skin and subcutaneous tissue disorders) | 98 | 103
Rash (Skin and subcutaneous tissue disorders) | 106 | 64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.